CLINICAL TRIAL: NCT05761418
Title: Preoperative Vaginal Dinoprostone Versus Misoprostone to Decrease Bleeding During Abdominal Myomectomy
Brief Title: Preoperative Vaginal Dinoprostone Versus Misoprostone in Abdominal Myomectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REC-H-PhBSU-22021
Record Dates: First submitted 2023-02-23; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Myoma;Uterus
Keywords: Uterine leiomyoma; misoprostol; dinoprostone
MeSH Terms: conditions — Myofibroma | interventions — Dinoprostone; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dinoprostone (Experimental): Will receive 20 mg of Dinoprostone vaginally 2 hrs. preoperatively.
  Interventions: Drug: Dinoprostone
- Misoprostol (Experimental): will receive 400 μg of Misoprostol vaginally 2 hrs. preoperatively.
  Interventions: Drug: Misoprostol
- control (No Intervention): received a placebo vaginally 2 hrs. preoperatively.

INTERVENTIONS:
Drug: Dinoprostone — prostaglandin (PG) E2 analog
  Other Names: Dinoglandin
  Arms: Dinoprostone
Drug: Misoprostol — prostaglandin (PG) E1 analog
  Other Names: Cytotec
  Arms: Misoprostol

SUMMARY:
Aim and objectives; To compare the efficacy of preoperative administration of dinoprostone 20 mg versus 400 ug misoprostol vaginally in decreasing the amount of bleeding during abdominal myomectomy

DETAILED DESCRIPTION:
Background; Myomectomy is a curative interventional option for many kinds of uterine fibroids, but considerable intraoperative haemorrhage and the necessities for transfusions of blood are still the main challenge for abdomen myomectomy.

Aim and objectives; To compare the efficacy of preoperative administration of dinoprostone 20 mg versus 400 ug misoprostol vaginally in decreasing the amount of bleeding during abdominal myomectomy Subjects and methods; This was a prospective randomized double-blind controlled study that included 90 patients complaining of uterine myoma and indicated for myomectomy selected from the outpatient clinic at Beni-suef university hospital

ELIGIBILITY:
Inclusion Criteria:

* Age 30-50 years
* all cases with uterine fibroid not responding to medical treatment and indicated for myomectomy.

Exclusion Criteria:

* contraindications to dinoprostone or misoprostol,
* active PID,
* history of pelvic/ ovarian endometriosis,
* females who had pre-operative mifepristone, GnRH analog or orally contraception drugs, earlier myomectomy.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Blood loss | all time of the myomectomy operation
  quantity of blood collected in the aspiration apparatus and the quantity of blood on the operative gauze.

SECONDARY OUTCOMES:
change hemoglobin levels | within 1 week before operation and 24 hours after operation
  Pre and Postoperative hemoglobin levels

CONTACTS AND LOCATIONS:
Overall Officials: Beni-Suef University, Principal Investigator — Faculty of Medicine Beni-Suef University
Locations (1):
- Beni-suef university, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No